CLINICAL TRIAL: NCT03974763
Title: Function and Form Outcomes in Patients With Facial Paralysis
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 11299
Record Dates: First submitted 2018-09-24; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Facial Paralysis; Bell Palsy
Keywords: Facial Paralysis; Bell's Palsy; unilateral; 3D; 3D imaging; Facial form; Facial function
MeSH Terms: conditions — Facial Paralysis; Bell Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Group: Patients with acute, unilateral, facial paralysis (Bell's Palsy)
- Control Group: A group of age- and sex-frequency matched 'normal' controls. Based on past research, gender and age are possible confounders of facial movement/function. Thus, the control group will be frequency-matched to the patient group on gender and age.

SUMMARY:
This study will be unique for the rehabilitation of patients with facial paralysis in that the focus is to generate novel 3D facial soft tissue measures to characterize the condition and temporal changes, and on the generation of future testable hypotheses to optimize surgical interventions and outcomes. In addition, the investigators will extend our previous work, beyond the facial circumoral and lip areas/zones, to characterize additional facial zones specific for facial paralysis.

The approach for facial mapping of soft tissue movement, when validated through this proposed study, can be used for both surgical planning and to support the development and training of implantable facial pacing devices. Mapping both normal facial movements and movements of patients with unilateral facial paralysis are vital to describe the temporal and spatial course of the recovery process. Ultimately, this information can be used to inform clinicians on the precise placement of these devices and the signal strength needed to facilitate movements in the required 'paralyzed' facial zones until the recovery process has been completed.

DETAILED DESCRIPTION:
Patients with facial paralysis have an obvious facial disability. The resultant facial disability includes facial disfigurement and impairment in soft tissue movements, particularly in facial expressive behaviors. These negative physical sequelae not only impact facial esthetics and function, but also patients' social and emotional quality of life. Treatments range from non-surgical interventions and facial reanimation surgery to new implantable facial pacing devices that would potentially initiate artificial movement on the paralyzed side of the face. Traditionally, surgeons' plan treatment based on isolated measurements made from 2D photographs and subjective grading of the patient's face, both of which are limited in scope and dimension. Our research group has demonstrated the utility of a novel 3D dynamic and static quantitative (objective) measures for the evaluation of facial soft tissue function. The measures are objective and quantitative, and they provide a more precise diagnosis of facial soft tissue disability and evaluation of surgical outcomes. The main goal of this prospective, observational study is to determine the applicability of these novel 3D dynamic and static measures for quantification and measurement of impairment and disfigurement, as well as change over time, in patients with facial paralysis. The global hypothesis is that the use of the measures will provide a more comprehensive analysis of the severity of facial paralysis and the changes over time (recovery) when compared with current assessment methods.

ELIGIBILITY:
Patients with Facial Paralysis Inclusion criteria

* A diagnosis of virally triggered, acute, unilateral facial paralysis (Bell's Palsy)
* Able to attend baseline visit at Tufts within 6 weeks of onset of the condition and with an estimated potential for recovery between 6-12 weeks
* Patient interest/willingness to participate in the study
* An ability to comprehend verbal instructions; and an age range of 18 to 75 years

Exclusion criteria

* Facial movement disorders due to primary muscular dysfunction or hemifacial spasm in the absence of synkinesis
* Complaints of facial paralysis but no evidence of weakness on physical examination
* Previous facial soft tissue surgery and/or Orthognathic surgery
* Mental or hearing impairment to the extent that comprehension or ability to perform the tests is hampered

Control Participants Inclusion criteria

* Subject interest/willingness to participate in the study
* An ability to comprehend verbal instructions
* An age range of 18 to 75 years

Exclusion criteria

* Facial soft tissue surgery, orthognathic surgery, and/or facial soft tissue disorder
* Mental or hearing impairment to the extent that comprehension or ability to perform the tests is hampered

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects for this study will be adults 18 to 75 years. The subjects who are potentially eligible for participation will be identified through the participating Centers: For the patients with facial paralysis through the Facial Nerve Center (FNC) at Massachusetts Eye and Ear Infirmary (MEEI); and for the control subjects through Tufts University School of Dental Medicine (TUSDM). Subjects recruited from MEEI will attend TUSDM for testing where Dr. Trotman maintains her Facial Animation laboratory. The participating surgeon is Dr. Tessa Hadlock and she will be responsible for the clinical care of all patients.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
To quantitatively evaluate the range of facial soft tissue disability in patients with acute, unilateral, flaccid facial paralysis and track the changes over time (3-month recovery period). | December 2019
  First outcome measure for facial soft tissue disability = Maximum displacement (mm)
To quantitatively evaluate the range of facial soft tissue disability in patients with acute, unilateral, flaccid facial paralysis and track the changes over time (3-month recovery period). | December 2019
  Second outcome measure for facial soft tissue disability = velocity (mm/s)
To quantitatively evaluate the range of facial soft tissue disability in patients with acute, unilateral, flaccid facial paralysis and track the changes over time (3-month recovery period). | December 2019
  Third outcome measure for facial soft tissue disability = and asymmetry of facial soft tissue landmarks (this is a ratio measure)
To compare the facial disability in the patients with a group of age- and sex-frequency matched normal subjects. | December 2019
  First outcome measure for group comparison = difference in maximum displacement (mm) between patients with facial disability and control group subjects
To compare the facial disability in the patients with a group of age- and sex-frequency matched normal subjects. | December 2019
  Second outcome measure for group comparison = velocity (mm/s)
To compare the facial disability in the patients with a group of age- and sex-frequency matched normal subjects. | December 2019
  Third outcome measure for group comparison = asymmetry of facial soft tissue landmarks (ratio)
In patients with acute, unilateral, flaccid facial paralysis, to compare the current, qualitative, clinical assessment methods for facial disability. | December 2019
  First outcome measure = average correlation across surgeons for their ratings on the House-Brackman scale and the patients' mean measures of maximum displacement
In patients with acute, unilateral, flaccid facial paralysis, to compare the current, qualitative, clinical assessment methods for facial disability. | December 2019
  Second outcome measure = average correlation across surgeons for their ratings on the House-Brackman scale and the patients' mean measures of velocity
In patients with acute, unilateral, flaccid facial paralysis, to compare the current, qualitative, clinical assessment methods for facial disability. | December 2019
  Third outcome measure = average correlation across surgeons for their ratings on the House-Brackman scale and the patients' mean measures of asymmetry of facial soft tissue landmarks
In patients with acute, unilateral, flaccid facial paralysis, to compare the current, qualitative, clinical assessment methods for facial disability. | December 2019
  Fourth outcome measure = average correlation across surgeons for their ratings on the Sunnybrook Facial Grading System and the patients' mean measures of maximum displacement
In patients with acute, unilateral, flaccid facial paralysis, to compare the current, qualitative, clinical assessment methods for facial disability. | December 2019
  Fifth outcome measure = average correlation across surgeons for their ratings on the Sunnybrook Facial Grading System and the patients' mean measures of velocity
In patients with acute, unilateral, flaccid facial paralysis, to compare the current, qualitative, clinical assessment methods for facial disability. | December 2019
  Sixth outcome measure = average correlation across surgeons for their ratings on the Sunnybrook Facial Grading System and the patients' mean measures of asymmetry of facial soft tissue landmarks
To assess perceptions of facial appearance over time in patients with acute, unilateral, flaccid facial paralysis and to compare these perceptions with those of control subjects. | December 2019
  Measurement Tools: SP36 questionnaire, FaCE questionnaire.
To assess perceptions of quality of life over time in patients with acute, unilateral, flaccid facial paralysis and to compare these perceptions with those of control subjects. | December 2019
  Measurement Tools: PSP questionnaire.
To correlate the patients' perceptions over time with the quantitative measures of facial disability. | December 2019
  Relationship between the quantitative measurements of facial movement with the quality of life and patient perception measures. This relationship will be measured using the linear mixed effects model or generalized estimating equations as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Carroll Ann Trotman, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States